CLINICAL TRIAL: NCT00799188
Title: CERTICOEUR a Secondary Prevention Study of Skin Cancers in Heart Transplant Patients. An Open Labelled Randomized Everolimus vs Calcineurin Inhibitors Multicenter Trial
Brief Title: CERTICOEUR: A Secondary Prevention Study of Skin Cancers in Heart Transplant Patients. Everolimus Versus Calcineurin Inhibitors Multicenter Trial
Acronym: CERTICOEUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007.489/32
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Transplantation; Skin Cancer
Keywords: Cardiac Transplantation; Skin cancer; Everolimus
MeSH Terms: conditions — Skin Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): reduction of immunosuppression
- 2 (Experimental): switch to Everolimus : 50% reduction of calcineurin inhibitors (ciclosporine or tacrolimus)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 50% reduction of calcineurin inhibitors daily dose followed by further decrease or withdrawal. Everolimus will be introduced and tapered to a trough level of 6 to 10 microg/l.
  Other Names: Certican
  Arms: 2

SUMMARY:
Heart transplant is a recognized therapeutic strategy in refractory heart failure. Its success is however hampered by severe cancer occurrence and recurrence. The new m-tor inhibiting drugs Sirolimus and Everolimus have shown potential for reducing the incidence of cancer in animal models. They are potent immunosuppressant, antiproliferative and antiangiogenic drugs. This open labelled randomized multicenter study aims at evaluating the beneficial antineoplastic effect of Everolimus in 159 heart transplant patients suffering of recurrent skin cancer. Primary objective is to demonstrate a reduction in the number of new skin cancers. Secondary end point will be time of recurrence, incidence of non skin cancer, graft function following switch (including death), renal function evolution following calcineurin inhibitors reduction or withdrawal, Everolimus tolerance profile, schemes of calcineurin inhibitors reduction management in centers.

DETAILED DESCRIPTION:
* Open labelled randomized Everolimus vs reduction of calcineurin inhibitors trial. 2:1 randomization design
* October 10, 2008
* 159 patients (106 everolimus vs 53 calcineurin inhibitors reduction)
* 175 patients (117 vs 58)
* X Not yet recruiting 0 recruiting 0 no longer recruiting
* Number of skin tumors per patients requiring surgery with histology control within 2 years

Within 2 years of Follow up:

* New skin cancer
* Number of patients with new skin cancers
* Time of recurrence
* Number and histology of other types of skin cancer
* Graft function (including acute rejection, graft loss, death)
* Renal function evolution as assessed using Cockcroft creatinine clearance and proteinuria
* Adverse events and serious adverse events
* Non skin cancer (Number and diagnostic)
* Schemes of calcineurin inhibitors reduction/withdrawal
* Immune response assessment through regulatory or effector function of blood and in situ T lymphocytes at baseline and following immunosuppression switch

ELIGIBILITY:
Inclusion Criteria:

* First orthotopic heart transplant after 1st year
* No rejection within previous 6 Months
* Occurrence of squamous cell carcinoma, basal cell carcinoma, in situ carcinoma, Bowen disease, premalignant keratosis
* Recurrence of skin cancers leading to immunosuppressive regimen modifications
* Removal of a skin lesion in the past three years
* Above 18 yrs and under contraceptive drugs if applicable
* Informed consent given
* Health coverage ongoing

Exclusion Criteria:

* Other non simultaneously transplanted organ
* recent biopsy proven acute rejection
* Proteinuria > 1g/l
* Ongoing infectious disease
* HIV positivity, Chronic active Hepatitis B or C.
* Abnormal blood tests: transaminases >= 3UNL, Bilirubin > 34 mmol.l, albumin<35 g/l, spontaneous INR >1,3
* Hemoglobin >= 8 g/dl, White Blood Count<= 2 giga/l, platelet count <= 50 giga/l
* Hypercholesterolemia>= 9 mmol/l, hypertriglyceridemia >= 8,5 mmol/l despite treatment
* History of macrolid or mTor inhibitor intolerance
* Previous cancer other than skin in the year prior to enrollment
* Medical or surgical condition unsuitable for the trial
* Breast feeding
* Positive pregnancy test
* Severe psychiatric disorder
* Communication or language disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-10; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of skin tumors per patients requiring surgery with histology control within 2 years | 2 years

SECONDARY OUTCOMES:
New skin cancer | 2 years
Number of patients with new skin cancers | 2 years
Time of recurrence | 2 years
Number and histology of other types of skin cancer | 2 years
Graft function (including acute rejection, graft loss, death) | 2 years
Renal function evolution as assessed using Cockcroft creatinine clearance and proteinuria | 2 years
Adverse events and serious adverse events | 2 years
Non skin cancer (Number and diagnostic) | 2 years
Schemes of calcineurin inhibitors reduction/withdrawal | 2 years
Immune response assessment through regulatory or effector function of blood and in situ T lymphocytes at baseline and following immunosuppression switch | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT SEBBAG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- HOSPICES CIVILS de LYON, Lyon, France